CLINICAL TRIAL: NCT02295839
Title: Feasibility, Acceptability, and Effectiveness of a Sleep Hygiene and Relaxation Intervention to Improve Sleep and Fatigue for Children Receiving Maintenance Chemotherapy for Acute Lymphoblastic Leukemia
Brief Title: Sleep Hygiene and Relaxation Intervention to Improve Sleep and Fatigue for Children Receiving Maintenance Chemotherapy
Acronym: SHARI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Sue Zupanec, Nurse Practitioner, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1000025162
Record Dates: First submitted 2014-11-17; First posted 2014-11-20 (Estimated); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Sleep; Fatigue; Acute Lymphoblastic Leukemia
Keywords: Sleep; Acute Lymphoblastic Leukemia; Fatigue; Sleep hygiene; Relaxation; RCT
MeSH Terms: conditions — Fatigue; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Sleep Hygiene

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (No Intervention)
- Sleep Hygiene and Relaxation Education (Experimental)
  Interventions: Behavioral: Sleep Hygiene and Relaxation Education

INTERVENTIONS:
Behavioral: Sleep Hygiene and Relaxation Education — Intervention group participants receive a nurse-led, one-hour 1:1 educational session including education about sleep in children and a description of what is known about sleep and fatigue issues in children with cancer. The session also includes strategies to improve sleep hygiene in children. Information about relaxation to promote sleep is outlined and two children's books designed to promote relaxation using the principles of deep breathing are given to the parent(s). A handout containing all the information covered is given to the parent(s).
  Arms: Sleep Hygiene and Relaxation Education

SUMMARY:
This pilot randomized controlled trial examined the feasibility, acceptability and effectiveness of an intervention to improve sleep quality and decrease fatigue levels in children with a diagnosis of ALL, during maintenance treatment. Families were randomized to usual care or the intervention. The intervention included a sleep hygiene and relaxation education session with a nurse practitioner, literature for home, two story books, and a follow-up phone call. Self-reported measures were used in addition to actigraphy to measure children's quality and quantity of sleep.

DETAILED DESCRIPTION:
Sleep is an essential restorative function that promotes both physical and cognitive health. Previous studies have demonstrated that children on Acute Lymphoblastic Leukemia (ALL) maintenance therapy have problematic sleep patterns and experience fatigue. This pilot randomized controlled trial examined the feasibility, acceptability and effectiveness of an intervention to improve sleep quality and decrease fatigue levels in children aged 4-10, with a diagnosis of ALL, during maintenance treatment. Families were randomized to usual care or the intervention. The intervention included a sleep hygiene and relaxation education session with a nurse practitioner, literature for home, two story books, and a follow-up phone call. Self-reported measures were used in addition to actigraphy to measure children's quality and quantity of sleep. Sleep tips were evaluated by intervention group families.

ELIGIBILITY:
Inclusion Criteria:

* Child aged 4-10 with a diagnosis of precursor acute B lymphoblastic leukemia (B ALL) in maintenance phase of therapy beyond 3rd course (protocol AALL0331)
* Child and parent able to understand and read English
* Child is within one year of age-appropriate grade in school

Exclusion Criteria:

* Child who is receiving palliative care
* Child with diagnosis of depression
* Child who has been prescribed medications for insomnia
* Child who has a physician-diagnosed sleep disorder (e.g. narcolepsy, restless legs syndrome)
* Child who has received radiation therapy
* Child has potential sleep disordered breathing (measured by Children's Sleep Habits Questionnaire)

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2011-05; Primary Completion 2013-06 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Feasibility and acceptability of intervention (The Evaluation of Sleep Tips form) | Weeks 1-4, post-intervention
  The Evaluation of Sleep Tips form will use open-ended questions to ask parents about factors that promoted or prevented implementing the sleep hygiene and relaxation interventions, and which components of the intervention they implemented and in what frequency.

SECONDARY OUTCOMES:
Nocturnal sleep (minutes) | Five consecutive nights on two occasions
  Sleep and wake times will be objectively collected using actigraphy.

OTHER OUTCOMES:
Sleep Disturbances (The Children's Sleep Habits Questionnaire) | Baseline, Weeks 4 and 8
  The Children's Sleep Habits Questionnaire will be used to measure usual sleep habits (sleep duration, consistency of sleep and wake times during the week, and between weekdays and weekends) as well as sleep problems in the most recent, typical week
School attendance | One month
  A calendar data form will be used by parents to mark if their child attended school for a full day, half day, or not at all. Reasons for absences will be collected.
Fatigue levels (Childhood Cancer Fatigue Scale-Child (FS-C) and the Childhood Cancer Fatigue Scale-Parent (FS-P) | Baseline, Weeks 4 and 8
  * Fatigue levels will be measure using the Childhood Cancer Fatigue Scale-Child (FS-C) and the Childhood Cancer Fatigue Scale-Parent (FS-P)
  * Children under the age of seven will not complete the FS-C
Daytime and pre-bedtime behaviours (The Family Inventory of Sleep Habits (FISH) | Baseline, Weeks 4 and 8
  The Family Inventory of Sleep Habits (FISH) will be used to measure daytime behaviours (e.g. exercise) and before bedtime behaviours (e.g. engaging in stimulating activity) known to influence sleep in children, along with the child's sleep environment and pre-bedtime routines.

CONTACTS AND LOCATIONS:
Overall Officials: Sue Zupanec, MN, NP-Peds, Principal Investigator — Hospital for Sick Children (SickKids)
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Result] Zupanec S, Jones H, McRae L, Papaconstantinou E, Weston J, Stremler R. A Sleep Hygiene and Relaxation Intervention for Children With Acute Lymphoblastic Leukemia: A Pilot Randomized Controlled Trial. Cancer Nurs. 2017 Nov/Dec;40(6):488-496. doi: 10.1097/NCC.0000000000000457. PMID 27922922